CLINICAL TRIAL: NCT03683875
Title: Ultrasonography of the Neuromuscular Degeneration Behavior in ALS: a Longitudinal Study
Brief Title: Ultrasonography of the Neuromuscular Degeneration Behavior in Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Santa Lucia (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio Tomás Ríos-Cortés, Msc Physiotherapist, Hospital General Universitario Santa Lucia
Other Study IDs: ECO-ELA
Record Dates: First submitted 2018-09-12; First posted 2018-09-25 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a progressive and fatal neurological disease.

An exhaustive and frequent clinical evaluation can lead to establish an adequate and early treatment of the consequences of its evolution.

Objectives.

1. To evaluate the evolution of diaphragmatic and peripheral neuromuscular degeneration by ultrasound examination in patients with ALS and to establish possible evolution patterns.
2. To verify the relationship between the degenerative peripheral and diaphragmatic neuromuscular changes evaluated by ultrasonography and changes in clinical scales frequently used.
3. To compare the ultrasonographic features of subjects with ALS and a sample of healthy subjects Methods. A longitudinal observational study in a consecutive sample of patients diagnosed with ALS will be realized. All the patients will be examined 3 times, with an interval of at least 3 months between tests. Bilateral and cross sectional ultrasonography of several peripheral muscles and diaphragm will be performed at rest and during muscle contraction. All the images will be processed and analyzed for obtaining morphometric variables (muscle thickness) and textural ones (echogenic variation, entropy, homogeneity, textural contrast and correlation). Frequency of twitches will be also recorded in peripheral muscles.Also clinical features will be noted, every time of the 3 exams, from Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-r), British Medical Council Research Scale(MRC), and routine pulmonary tests.

ELIGIBILITY:
Inclusion Criteria:

* Definite ALS

Exclusion Criteria:

* Primary Lateral Sclerosis (PLS)
* Other forms of motor neuron disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Amyotrophic Lateral Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Measuring thickness of peripheral muscles using an ultrasound device | 3 months
  These measurements will be carried out in the biceps brachialis, forearm flexors, thenar eminence muscle, quadriceps and tibialis anterior which will be compared between patient with ALS and control group.
Measuring echointensity of peripheral muscles using an ultrasound device | 3 months
  These measurements will be carried out in the biceps brachialis, forearm flexors, thenar eminence muscle, quadriceps and tibialis anterior which will be compared between patient with ALS and control group.
Measuring sonoelastography of peripheral muscles using an ultrasound device | 3 months
  These measurements will be carried out in the biceps brachialis, forearm flexors, thenar eminence muscle, quadriceps and tibialis anterior which will be compared between patient with ALS and control group.
Thickness Fraction of the Diaphragm in ALS patients and control group. | 3 months
  It is calculated as the difference between thickness at end inspiration and end expiration
Diaphragmatic Excursion (quiet and forced) of the Diaphragm in ALS patients and control group | 3 months
  Displacement of the right diaphragm dome

SECONDARY OUTCOMES:
Measurement of muscle fasciculations using an ultrasound device | 3 months
  Each peripheral muscle will be screened during 30 seconds
Measurement of muscle strength using Medical Research Council Scale (MRCs) | 3 months
  Graded on the medical research council scale. This scale grades muscle power on a scale of 0 to 5:
  Grade 0: no movement is observed Grade 1: only a trace or flicker of movement is seen or flet in the muscle. or fasciculation is observed Grade 2: movement is possible only if the resistance of gravity is removed Grade 3: movement against gravity is possible but not against resistance of the examiner Grade 4: muscle stregth is reduced but muscle contraction can move joint against gravity and resistance Grade 5: muscle contracts normally against full resistance
Measurement Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-r) | 3 months
  Questionnaire with 12 items with a score from 0 to 4 each item:
  1. Speech
  2. Salivation
  3. Swallowing
  4. Handwriting 5a. Cutting food and handling utensils (patients without gastrostomy) 5b. Cutting food and handling utensils(scale for patients with gastrostomy)
  6. Dressing and hygiene 7. Turning in bed and adjusting bed clothes 8. Walking 9. Climbing stairs 10. Dyspnea 11. Orthopnea 12. Respiratory insufficiency
  There are three main pathways of progression, the questions are also divided in relation to the types of onset. Questions 1 to 3 are related to bulbar onset, questions 4 to 9 are related to limb onset and questions 10-12 are related to respiratory onset. The Scale goes from 0 to 48, more points meaning better situation.
Measuring Forced Vital Capacity | 3 months
  This volume expressed in liters will be measured in supine and seated positions.
Maximal Inspiratory Pressure (MIP) | 3 months
  Measure of the strength of inspiratory muscles expressed in centimeters of water, is the highest mouth pressure sustained for 1 s during a maximum inspiratory effort
Sniff- nasal inspiratory pressure (SNIP) | 3 months
  It consists of measuring nasal pressure in an occluded nostril during a maximal sniff performed through the contralateral nostril, expressed in centimeters of water
Peak Cough Flow (PCF) | 3 months
  Maximal peak cough flow expressed in liters per minute
Partial Pressure of Carbon Dioxide in Arterial Blood (PaCO2) | 3 months
  Obtained by a radial arterial blood sample and expressed in millimeters of mercury
Cumulative time percentage with SpO2 under 90% (CT90) | 3 months
  SpO2 is an estimate of arterial oxygen saturation expressed in percentage under 90% obtained from a nocturnal oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Tomás Ríos Cortés, Principal Investigator — HOSPITAL GENERAL UNIVERSITARIO SANTA LUCIA - SERVICIO MURCIANO DE SALUD
Locations (1):
- Hospital General Universitario Santa Lucia, Cartagena, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayans D, Cartwright MS, Walker FO. Neuromuscular ultrasonography: quantifying muscle and nerve measurements. Phys Med Rehabil Clin N Am. 2012 Feb;23(1):133-48, xii. doi: 10.1016/j.pmr.2011.11.009. Epub 2011 Dec 9. PMID 22239880
- [Background] Arts IMP, Overeem S, Pillen S, Jurgen Schelhaas H, Zwarts MJ. Muscle changes in amyotrophic lateral sclerosis: a longitudinal ultrasonography study. Clin Neurophysiol. 2011 Mar;122(3):623-628. doi: 10.1016/j.clinph.2010.07.023. PMID 20810308
- [Background] Arts IM, Overeem S, Pillen S, Kleine BU, Boekestein WA, Zwarts MJ, Jurgen Schelhaas H. Muscle ultrasonography: a diagnostic tool for amyotrophic lateral sclerosis. Clin Neurophysiol. 2012 Aug;123(8):1662-7. doi: 10.1016/j.clinph.2011.11.262. Epub 2012 Jan 13. PMID 22244867
- [Background] Arts IM, Overeem S, Pillen S, Schelhaas HJ, Zwarts MJ. Muscle ultrasonography to predict survival in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2011 May;82(5):552-4. doi: 10.1136/jnnp.2009.200519. Epub 2010 Apr 14. PMID 20392981
- [Background] Arts IM, van Rooij FG, Overeem S, Pillen S, Janssen HM, Schelhaas HJ, Zwarts MJ. Quantitative muscle ultrasonography in amyotrophic lateral sclerosis. Ultrasound Med Biol. 2008 Mar;34(3):354-61. doi: 10.1016/j.ultrasmedbio.2007.08.013. Epub 2007 Oct 26. PMID 17964067
- [Background] Arts IM, Pillen S, Schelhaas HJ, Overeem S, Zwarts MJ. Normal values for quantitative muscle ultrasonography in adults. Muscle Nerve. 2010 Jan;41(1):32-41. doi: 10.1002/mus.21458. PMID 19722256
- [Background] Schreiber S, Abdulla S, Debska-Vielhaber G, Machts J, Dannhardt-Stieger V, Feistner H, Oldag A, Goertler M, Petri S, Kollewe K, Kropf S, Schreiber F, Heinze HJ, Dengler R, Nestor PJ, Vielhaber S. Peripheral nerve ultrasound in amyotrophic lateral sclerosis phenotypes. Muscle Nerve. 2015 May;51(5):669-75. doi: 10.1002/mus.24431. Epub 2015 Mar 14. PMID 25155020
- [Background] Cartwright MS, Walker FO, Griffin LP, Caress JB. Peripheral nerve and muscle ultrasound in amyotrophic lateral sclerosis. Muscle Nerve. 2011 Sep;44(3):346-51. doi: 10.1002/mus.22035. Epub 2011 Aug 3. PMID 21815172
- [Background] Martinez-Paya JJ, Del Bano-Aledo ME, Rios-Diaz J, Tembl-Ferrairo JI, Vazquez-Costa JF, Medina-Mirapeix F. Muscular Echovariation: A New Biomarker in Amyotrophic Lateral Sclerosis. Ultrasound Med Biol. 2017 Jun;43(6):1153-1162. doi: 10.1016/j.ultrasmedbio.2017.02.002. Epub 2017 Apr 8. PMID 28395965
- [Background] Martinez-Paya JJ, Rios-Diaz J, Del Bano-Aledo ME, Tembl-Ferrairo JI, Vazquez-Costa JF, Medina-Mirapeix F. Quantitative Muscle Ultrasonography Using Textural Analysis in Amyotrophic Lateral Sclerosis. Ultrason Imaging. 2017 Nov;39(6):357-368. doi: 10.1177/0161734617711370. Epub 2017 May 28. PMID 28553752
- [Background] Hiwatani Y, Sakata M, Miwa H. Ultrasonography of the diaphragm in amyotrophic lateral sclerosis: clinical significance in assessment of respiratory functions. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Mar;14(2):127-31. doi: 10.3109/17482968.2012.729595. Epub 2012 Oct 30. PMID 23110443
- [Background] Pinto S, Alves P, Pimentel B, Swash M, de Carvalho M. Ultrasound for assessment of diaphragm in ALS. Clin Neurophysiol. 2016 Jan;127(1):892-897. doi: 10.1016/j.clinph.2015.03.024. Epub 2015 Apr 25. PMID 25971723
- [Background] Fantini R, Mandrioli J, Zona S, Antenora F, Iattoni A, Monelli M, Fini N, Tonelli R, Clini E, Marchioni A. Ultrasound assessment of diaphragmatic function in patients with amyotrophic lateral sclerosis. Respirology. 2016 Jul;21(5):932-8. doi: 10.1111/resp.12759. Epub 2016 Mar 19. PMID 26994409